CLINICAL TRIAL: NCT06077851
Title: Continuous Monitoring With Real-time Transmission of Vital Signs to Healthcare Professionals From Patients at Home
Brief Title: Continuous Monitoring of Vital Signs at Home (WARD HOME II)
Status: Recruiting | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Technical University of Denmark (Other); Emergency Medical Services, Capital Region, Denmark (Other Government)
Responsible Party: Principal Investigator, Emilie Sigvardt, Principal investigator, Bispebjerg Hospital
Other Study IDs: 2308603
Record Dates: First submitted 2023-09-27; First posted 2023-10-11 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-06

CONDITIONS: Vital Sign Monitoring; Clinical Deterioration; Hospital At Home
MeSH Terms: conditions — Clinical Deterioration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Continuously monitoring — Included patients are monitored with WARD equipment the first days after discharge. Monitoring will last for a maximum of three days.

SUMMARY:
The study aims to investigate the use of wireless, continuous monitoring in patients at home including the frequency of alarms triggered by abnormal vital parameters and their significance for (re)hospitalisation/Serious Adverse Events(SAE) and/or death within 30 days.

DETAILED DESCRIPTION:
Acute hospital admissions challenge the capacity of the healthcare system. Readmission is common among patients with chronic medical diseases, and many patients admitted for acute conditions are often subsequently observed at the hospital for hours and often with one overnight stay for observation purposes alone. Recent medico technical research has allowed continuous and wireless monitoring of patients' vital signs in-hospital, but the practice at home remains uninvestigated. However, the technology has the potential to relieve hospital overcrowding by offering continuous and real time analytics of vital signs in high-risk patients at home.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (≥18 years) admitted (with at least one night stay) with an acute medical disease and scheduled for discharge to their own homes

Adult patients (≥18 years) who have contacted the EMS and, after assessment by paramedic personnel, not deemed sick enough for immediate hospital admission.

Exclusion Criteria:

Patients placed on palliative treatment.

Acceptable chronically abnormal vital parameters of SpO2<88%, MAP<70, RR>24, or HR>110.

Allergy to plaster, plastic, or silicone.

A pacemaker or Implantable Cardioverter Defibrillator (ICD) device.

If the patient was deemed not able to open the front door when visited by the investigator.

Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with an acute medical disease at Bispebjerg Hospital or Rigshospitalet, or assessed by paramedic personnel at home after contact to the EMS.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
(Re)admission | within 30 days
  Defined as acute admission to hospital for at least 12 hours with relation to prior discharge or EMS contact
Serious Adverse Events | within 30 days
  Any adverse event, including acute admissions during the observational period. Criteria defined in protocol. Adverse events will be manually categorised as a 'severe adverse event' (SAE), or simple 'adverse event' (AE).
Mortality | within 30 days

SECONDARY OUTCOMES:
(Re)admission | within 7 days after discharge/assessment by paramedic personnel
  Defined as acute admission to hospital for at least 12 hours with relation to prior discharge or EMS contact
Inquiries to the Emergency Medical Service | within 30 days
  Defined as patients calls to 1813/112
Mortality and types of SAEs | within 30 days
  Any adverse event, including acute admissions during the observational period. Criteria defined in protocol. Adverse events will be manually categorised as a 'severe adverse event' (SAE), or simple 'adverse event' (AE).

OTHER OUTCOMES:
Frequency of automatically generated alerts on deviating vital signs | 72 hours
  per device per patient per day
Number of automatically generated alerts | 72 hours
  From all devices worn, per patient per day
Frequency of alerts which are responded to by healthcare personnel | 72 hours
  Number of alerts triggered by deviating vital signs, per patient per day
Fraction of time within the study period with at least one type of data transmitted in real time from patients' homes. | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Sigvardt, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, NV, Denmark

IPD SHARING:
Plan to Share IPD: Undecided